CLINICAL TRIAL: NCT05700799
Title: HEalth Advocate for Liver Transplant - Pilot
Acronym: HEAL-Tx Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-36504; K23DK132454 (NIH)
Record Dates: First submitted 2023-01-05; First posted 2023-01-26 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Liver Transplant; Complications; Pediatric ALL
Keywords: Health Advocate; Patient Navigator
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Patient Navigation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): This is a single arm pilot intervention.
  Interventions: Behavioral: Health Advocate

INTERVENTIONS:
Behavioral: Health Advocate — The Health Advocate intervention will include helping pediatric liver transplant recipients and their families address unmet household social needs (e.g., food insecurity), improve patient-provider communication, and enhance care coordination.
  Other Names: Patient Navigator

SUMMARY:
The Health Advocate for Liver Transplant (HEAL-Tx) Pilot is a nonrandomized, open-label intervention pilot of a health advocate intervention aimed to assess feasibility and acceptability of integrating a Health Advocate onto the transplant team. Across studies, health advocate roles vary, and can include coordinating medical care treatment, facilitating financial assistance (e.g., taxi vouchers), and connecting patients to community resources, which can improve self-management, mitigate social risks, and lead to better communication between the healthcare system and the family. In this pilot, the investigators will adapt this intervention for pediatric liver transplant patients and measure acceptability and feasibility according to RE-AIM.

ELIGIBILITY:
Inclusion Criteria:

1. Patients under 18 years if age that have undergone liver transplantation.
2. Subject and/or parent/legal guardian can provide written informed consent and willing to comply with study procedures.
3. Subject and/or parent/ legal guardian is willing to be contacted in the future by study staff.
4. Patient and/or caregiver felt to be a good fit for this pilot by transplant team.

Exclusion Criteria:

* Caregiver unwilling or unable to complete the survey.
* Child is a ward of the state (e.g. foster care) since present circumstances may not be reflective of child's past or future circumstances.
* Non-English, non-Spanish speakers.
* Non-US residents.
* Greater than 18 years of age at the time of enrollment.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in caregiver experience | Baseline and 90 days
  The investigators will administer a survey of caregiver experiences at study enrollment and at the end of the intervention to assess for changes in caregiver experience with the transplant team. These questions will focus on experiences receiving transplant care, experiences discussing social needs with the transplant team, and overall caregiver subjective assessment of the transplant recipient's overall health.

SECONDARY OUTCOMES:
Change in medication adherence using MLVI | Baseline, 90 days, and 180 days
  Medication level variability index (MLVI) defined as the standard deviation of 3 outpatient tacrolimus trough levels (binary >/=2.0 or <2.0). The investigators will assess this at study entry, intervention completion, and 6 months after study entry.
The quality of health advocate interactions with the participants, healthcare team, and community-based resources. | 90 days
  The Health Advocate will keep a detailed journal entry after each encounter and certain Health Advocate interactions will be recorded. The investigators will qualitatively analyze these journal entries and recordings to identify what functions the health advocate undertook.
A qualitative assessment of caregiver and healthcare provider satisfaction with the Health Advocate intervention. | 90 days
  The investigators will conduct in-depth interviews with the caregiver participant and clinical team members to assess overall satisfaction with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sharad Wadhwani, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No